CLINICAL TRIAL: NCT07201129
Title: A Phase 3, Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel-group Trial to Assess the Efficacy, Safety and Tolerability of Cenerimod in Adult Patients With Systemic Lupus Erythematosus and Active Lupus Nephritis in Combination With Background Therapy
Brief Title: A Research Trial to Assess if Cenerimod is Efficacious and Safe to Treat Active Lupus Nephritis on Top of Regular Treatment
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Viatris Innovation GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID-064B301
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-09

CONDITIONS: Nephritis, Lupus; Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic | interventions — cenerimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cenerimod 4 mg (Experimental): Participants will receive cenerimod once daily in addition to background lupus nephritis (LN) therapy.
  Interventions: Drug: Cenerimod
- Matching placebo (Placebo Comparator): Participants will receive matching placebo once daily in addition to background LN therapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cenerimod — Cenerimod will be supplied as a film-coated tablets at the dose of 4 mg.
  Other Names: ACT-334441
  Arms: Cenerimod 4 mg
Drug: Placebo — Matching placebo will be supplied as identical film-coated tablets formulated with the same excipients but without the active ingredient, cenerimod.
  Arms: Matching placebo

SUMMARY:
The goal of this clinical trial is to learn if cenerimod, on top of regular treatment, works to treat active lupus nephritis in adults with systemic lupus erythematosus and active lupus nephritis. It will also learn about the safety of cenerimod. The main questions it aims to answer are:

* Does cenerimod improve kidney function in participants?
* What medical problems do participants have when taking cenerimod?

Researchers will compare cenerimod to a placebo (a look-alike substance that contains no drug) to see how well cenerimod works when it is added to regular treatment.

Participants will:

* Take cenerimod or a placebo every day for 76 weeks (approximately 1.5 years), on top of regular treatment.
* Visit the clinic every 1 to 3 months for checkups and tests.

ELIGIBILITY:
Main Inclusion Criteria:

* Classification of systemic lupus erythematosus (SLE) made according to the 2019 European Alliance of Associations for Rheumatology / American College of Rheumatology (EULAR/ACR) criteria.
* Renal biopsy within 6 months prior to Screening visit indicating Class III or IV active glomerulonephritis with or without co-existing Class V, OR pure Class V membranous LN. If no biopsy was performed within 6 months of Screening, a biopsy will be performed during the Screening period, after all other inclusion/exclusion criteria are verified.
* Active renal disease defined as urine protein/creatinine ratio ≥ 1 mg/mg, assessed on a 24h urine collection.
* eGFR ≥ 15 mL/min/1.73 m^2. Enrollment of participants with eGFR between ≥ 15 and < 30 mL/min/1.73 m^2 requires:

  * a renal biopsy during the screening period showing sclerosis in ≤ 50% of glomeruli,
  * activity index ≥ 2, and chronicity index < 4, on the National Institutes for Health 2018 activity and chronicity indices. These indices must be assessed on the kidney biopsy dated less than 6 months prior to Screening and confirmed by a nephropathologist.
* Initiation of the induction therapy with the mandatory following background therapy:

  1. Mycophenolate mofetil 1-3 g/day orally or mycophenolate sodium 720-2160 mg/day orally at Randomization. This treatment can be in place before Screening or started at Screening.
  2. Corticosteroids: 1-3 intravenous (i.v.) pulses of methylprednisolone at 250 to 1000 mg/pulse/day (maximum cumulative 3000 mg) followed by oral prednisone (or equivalent) at 0.5 mg/kg/day with a cap at 40 mg/day. Pulses can be administered during screening and up to 2 weeks prior to screening. Participants who cannot take the pulse i.v. corticosteroid therapy should directly start on 0.8-1.0 mg/kg/day (max 80 mg/day) oral prednisone (or equivalent), within the same window as i.v. pulses.

Note: If treatment with an antimalarial or belimumab is taken, it must be initiated at least 4 weeks prior to Screening and must be at stable dose during these 28 days prior to Randomization and continued at a stable dose until End-of-Treatment. Participants on azathioprine must be switched to mycophenolate mofetil or mycophenolate sodium prior to Randomization.

* Participants of childbearing potential must agree to:

  * Use a highly effective method of contraception from Visit 1 up to at least 24 weeks after discontinuation of trial intervention.
  * Undertake monthly urine pregnancy tests during the trial and up to at least 24 weeks after discontinuation of trial intervention.

Main Exclusion Criteria:

* Severe active central nervous system lupus
* History of, or current renal diseases (other than LN) that, in the opinion of the investigator, could interfere with the LN assessment and confound the disease activity assessment (e.g., diabetic nephropathy), or require dialysis, transplantation or end-stage renal disease.
* History or presence of Mobitz type II or third-degree atrioventricular block, sick sinus syndrome, symptomatic bradycardia, or syncope associated with cardiac disorders.
* Participants who experienced myocardial infarction, unstable angina pectoris, stroke, transient ischemic attack, vascular thrombosis, decompensated heart failure requiring hospitalization, or heart failure defined by the New York Heart Association Class III/IV within 6 months prior to Screening.
* Resting heart rate < 50 bpm as measured by the 12-lead electrocardiogram (ECG) at Screening or at Randomization.
* Diagnosis of active or latent tuberculosis at Screening or within 6 months prior to Screening
* Negative antibody test for varicella-zoster virus
* Positive results for serological markers for hepatitis A, B, C and E indicating acute or chronic infection
* Participants with a positive human immunodeficiency virus (HIV) test or who have any other congenital or acquired immunodeficiency
* Presence of any of the following abnormalities, detected during the ophthalmological evaluation and/or by optical coherence tomography, as evaluated by the site ophthalmologist, during Screening:

  * Macular edema of any cause: diabetic, cystoid, tractional.
  * Foveal degeneration: macular hole, macular pseudohole, hereditary or degenerative maculopathies.
  * Active uveitis, papilledema.
  * Retinal neovascularization of any cause and in any location.
* Significant hematology abnormality at Screening:

  * Hemoglobin < 7 g/dL;
  * Lymphocyte count < 500 /μL (0.5 × 10^9/L);
  * White blood cell count < 1500/μL (1.5 × 10^9/L) or
  * Platelets < 25,000/μL (25 × 10^9/L)
* Treatment with the following medications within 5 half-lives of the medication prior to Randomization: Cyclosporine, voclosporin, tacrolimus, sirolimus, cyclophosphamide.
* Treatment with the following medications within 90 days prior to Randomization:

  * Leflunomide.
  * i.v. immunoglobulins.
  * Methotrexate.
  * Tyrosine kinase inhibitors.
* Treatment with anifrolumab within 6 months prior to Randomization.
* Treatment with biological immunosuppressive agents, (e.g., anti-tumor necrosis factor [anti-TNF], anti-interleukin-1 [anti-IL1], anti-IL6 therapies) within 90 days prior to Randomization.
* Treatment with B cell-depleting biological agents (e.g., rituximab, obinutuzumab or ocrelizumab) within 12 months prior to Randomization.
* Treatment with any of the following medications any time prior to Screening:

  * Alemtuzumab.
  * Sphingosine-1-phosphate receptor modulators (e.g., fingolimod).
  * Participants previously randomized to cenerimod or placebo in any trial involving cenerimod.
* Pregnancy confirmed via a serum pregnancy test at Visit 1 or a urine/serum pregnancy test at Visit 2 or planning to become pregnant, or lactating participant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-08 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Complete renal response (CRR) | At Week 76
  CRR at Week 76, defined as (both must be met):
  * Urine protein to creatinine ratio (UPCR) ≤ 0.5 mg/mg AND
  * No decrease from baseline of ≥ 20% in estimated glomerular filtration rate (eGFR)

SECONDARY OUTCOMES:
CRR while maintaining a low dose of corticosteroids | At Week 76
  • CRR at Week 76 with oral daily dose of 5 mg/day prednisone equivalent or less from Week 24 onwards
Time from randomization to sustained CRR | From Randomization to Week 76
  • Time from randomization to sustained CRR. Sustained CRR is defined as CRR criteria met for 2 consecutive visits.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Viatris Innovation GmbH
Locations (1):
- Allied Biomedical Research Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No